CLINICAL TRIAL: NCT05585554
Title: Locally Advanced Pancreatic Cancer Treated With ABLAtivE Stereotactic MRI-guided Adaptive Radiation Therapy (LAP-ABLATE)
Brief Title: Locally Advanced Pancreatic Cancer Treated With ABLAtivE Stereotactic MRI-guided Adaptive Radiation Therapy
Acronym: LAP-ABLATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAP-ABLATE
Record Dates: First submitted 2022-10-10; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
Keywords: Locally Advanced Pancreatic Cancer; SBRT; Radiation Therapy; MRIdian; ViewRay
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ablative MRIdian SMART (Experimental): Induction Chemotherapy + MRIdian SMART 50 Gy in 5 fractions
  Interventions: Radiation: MRIdian
- No ablative MRIdian SMART (No Intervention): Induction chemotherapy alone

INTERVENTIONS:
Radiation: MRIdian — Stereotactic MRI-guided On-table Adaptive Radiation Therapy delivered on MRIdian linac
  Arms: Ablative MRIdian SMART

SUMMARY:
Ablative dose magnetic resonance imaging (MRI) guided hypofractionated radiation therapy delivered using daily adaptive dose planning has shown to improve overall survival, relative to patients receiving lower radiation doses, in patients with locally advanced pancreatic cancer, without increasing the rate of serious gastrointestinal toxicity. The next step is to determine how these results compare to chemotherapy alone.

This is a prospective, randomized controlled trial (2:1) comparing induction chemotherapy followed by ablative Stereotactic MR-guided on-table Adaptive Radiation Therapy (SMART) versus chemotherapy alone in locally advanced pancreatic cancer patients. Overall survival outcomes at 2-years will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced pancreatic adenocarcinoma or adenosquamous carcinoma as defined by NCCN guidelines.
2. Minimum of 4 months interval from chemotherapy start to administration of the last dose/chemo.
3. Minimum 8 cycles of (m)FOLFIRINOX OR 12 doses of gemcitabine/nab - paclitaxel)
4. No radiographic evidence of local or distant disease progression at any time prior to study enrollment after starting chemotherapy
5. At least 18 years of age
6. ECOG performance status ≤ 1
7. Adequate bone marrow and organ function as defined below:

   1. Absolute neutrophil count ≥ 1,000/mcL
   2. Platelets ≥ 75,000/mcL
   3. Hemoglobin ≥ 8.0 g/dL
   4. Total bilirubin ≤ 1.5 x IULN
   5. AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
8. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
9. Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

1. CA19-9 > 180 U/mL within 30 days of randomization.
2. Any prior abdominal radiation therapy.
3. History of prior malignancy with the exception of: 1) malignancy treated with curative intent and with no known disease for at least 2 years from treatment to study enrollment, 2) adequately treated carcinoma in situ without evidence of disease (i.e. superficial bladder cancer).
4. Currently receiving any other investigational agents.
5. More than one cytotoxic regimen given for pancreatic cancer.
6. Major abdominal surgery within 4 weeks prior to randomization.
7. Definitive surgery for pancreas cancer completed prior to study enrollment (e.g., Whipple procedure).
8. Subject with planned or scheduled definitive surgery for pancreas at time of study enrollment
9. Grade 3 or greater toxicity during induction chemotherapy that has not resolved to at least grade 2
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
11. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
12. Medical/psychological contraindication to having an MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2-years
  To demonstrate superior 2-year overall survival from date of randomization in ablative MRIdian SMART versus no ablative MRIdian SMART in locally advanced pancreatic cancer patients without disease progression after induction chemotherapy.
  A Kaplan-Meier survival curve will be used to report the fraction of subjects living throughout the study

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2-years
  To demonstrate superior progression-free survival at 2 years from date of randomization in ablative MRIdian SMART therapy versus no ablative MRIdian SMART therapy in locally advanced pancreatic cancer patients without disease progression after induction chemotherapy.
  A Kaplan-Meier survival curve will be used to report percentage of patients living with pancreatic cancer without disease progression
Local Control (LC) | 2-years
  To compare local control at 2 years from date of randomization in ablative MRIdian SMART therapy versus no ablative MRIdian SMART therapy in locally advanced pancreatic cancer patients without disease progression after induction chemotherapy.
  A Kaplan-Meier curve will be used to report percentage of patients with local control of pancreatic cancer
Regional Control (RC) | 2-years
  To compare regional control at 2 years from date of randomization in ablative MRIdian SMART therapy versus no ablative MRIdian SMART therapy in locally advanced pancreatic cancer patients without disease progression after induction chemotherapy.
  A Kaplan-Meier curve will be used to report percentage of patients with regional control of pancreatic cancer
Distant Metastasis Free Survival (DMFS) | 2-years
  To compare distant metastasis free survival at 2 years from date of randomization in ablative MRIdian SMART therapy versus no ablative MRIdian SMART therapy locally advanced pancreatic cancer patients without disease progression after induction chemotherapy
  A Kaplan-Meier survival curve will be used to report percentage of patients living with pancreatic cancer without distant metastasis
Patient Reported Quality of Life (QoL) using EORTC QLQ-C30 questionnaire | 3-months, 12-months, 24-months
  To determine changes in patient-reported quality of life in patients diagnosed with locally advanced pancreatic cancer randomized post-chemotherapy with no disease progression in both study groups.
  The EORTC QLQ-C30 Scoring Manual will be followed for scoring.
  The QLQ-C30 consists of 28 four-level Likert items (on a scale of 1 - "Not at all" to 4 - "Very much"), and two seven-level Likert items which are scored according to the EORTC scoring guidelines into the 15 domains (Overall health and quality of life on a scale of 1 - "Very Poor" to "7 - Excellent").
  High scores in the 28 four-level Likert items indicate worse symptoms and health related QoL.
  High scores in the two seven-level Likert items indicate better health and quality of life related QoL.
Patient Reported Quality of Life (QoL) using EORTC QLQ-PAN26 questionnaire | 3-months, 12-months, 24-months
  To determine changes in patient-reported quality of life in patients diagnosed with locally advanced pancreatic cancer randomized post-chemotherapy with no disease progression in both study groups.
  The EORTC QLQ-C30 Scoring Manual will be followed for the supplemental QLQ-PAN26 module.
  The QLQ-PAN26 consists of 26 four-level Likert items (on a scale of 1 - "Not at all" to 4 - "Very much") which are scored according to draft scoring procedures supplied by EORTC to obtain seven multi-item scale scores consisting of two to four items and nine single-item scores.
  Higher scores indicate worse symptoms, function and health related QoL.
Treatment-related toxicity | 90 days
  To evaluate acute grade 3 or greater treatment-related toxicity (assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5) from randomization in patients diagnosed with locally advanced pancreatic cancer randomized post-chemotherapy with no disease progression in both study groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudra S, Jiang N, Rosenberg SA, Olsen JR, Roach MC, Wan L, Portelance L, Mellon EA, Bruynzeel A, Lagerwaard F, Bassetti MF, Parikh PJ, Lee PP. Using adaptive magnetic resonance image-guided radiation therapy for treatment of inoperable pancreatic cancer. Cancer Med. 2019 May;8(5):2123-2132. doi: 10.1002/cam4.2100. Epub 2019 Apr 1. PMID 30932367
- [Background] Eaton AA, Karanicolas P, Johnson MChir CD, Bottomley A, Allen PJ, Gonen M. Psychometric Validation of the EORTC QLQ-PAN26 Pancreatic Cancer Module for Assessing Health Related Quality of Life after Pancreatic Resection. JOP. J Pancreas (Online) 2017; 18(1):19-25.